CLINICAL TRIAL: NCT01220895
Title: A Prospective Phase II Study to Investigate the Efficacy and Safety of Pre-emptive Cytomegalovirus Adoptive Cellular Therapy in Patients Receiving Allogeneic Haematopoietic Stem Cell Transplant From an Unrelated Donor
Brief Title: Alternate Donor Study of Pre-Emptive Cellular Therapy
Acronym: CMV-ACE/ASPECT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cell Medica Ltd (Industry)
Collaborators: Leukaemia Lymphoma Research (Other); National Health Service, Blood and Transplant (Unknown); University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CM-2009-01
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Cytomegalovirus Infection
Keywords: Adoptive cellular therapy; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACT (mutlimer selection) plus standard therapy (Experimental): Adoptive Cellular Therapy prepared using Multimer Selection in combination with standard best available antiviral drug therapy
  Interventions: Biological: CMV-specific T-cells, single infusion following single positive CMV PCR result
- Best available antiviral drug therapy (Active Comparator)
  Interventions: Biological: CMV-specific T-cells, single infusion following single positive CMV PCR result

INTERVENTIONS:
Biological: CMV-specific T-cells, single infusion following single positive CMV PCR result — 1. Intravenous ganciclovir 5mg/kg twice daily
  2. Oral valganciclovir 900mg twice daily
  3. Intravenous foscarnet 90 mg/kg twice daily

SUMMARY:
The purpose of this study is to evaluate the potential clinical benefit of pre-emptive cytomegalovirus (CMV)-specific adoptive cellular therapy following T cell depleted allogeneic hematopoietic stem cell transplantation (HSCT) for reducing recurrent CMV reactivation.

DETAILED DESCRIPTION:
As with other herpes viruses, infection with CMV is thought to result primarily from reactivation of latent virus. Transmission of the virus can also occur from donor marrow infusion or from allogeneic red cell, leukocyte or platelet transfusions. However, in immunocompromised bone marrow transplant recipients, CMV is frequently reactivated and disease resulting from the progression of CMV infection is a major cause of infectious morbidity and mortality. CMV infection is a consequence both of the immunosuppression these patients receive and also may reflect delayed immune reconstitution in these patients following transplant. It is of particular concern to recipients of VUD (HLA-Volunteer Unrelated Donor) transplants who often receive lower doses of donor T cells in the transplant and who also require greater post-transplant immunosuppression for GVHD prophylaxis. CMV reactivation is most frequent in this group of transplant recipient.

One approach to improve reconstitution of immunity against viruses following allogeneic HSCT is to adoptively transfer donor-derived virus-specific T lymphocytes, which has been well documented with proven success. Existing evidence suggests that adoptive cellular therapy (ACT) can be an effective approach for treating viral reactivation following allo HSCT, with a minimal risk of inducing GVHD. The major advantage to the patient is likely to be avoidance of extended periods of therapy with antiviral medications that have significant associated morbidities, and sometimes require inpatient care. From a pharmacoeconomic viewpoint this would translate into a reduction of costs associated with standard antiviral therapies compared to the cost of adoptive cellular therapy.

It is anticipated that the use of very small numbers of highly specific T-cells will allow enough CMV-specific T-cells to be obtained in vitro from normal healthy CMV-seropositive donors from the peripheral blood transplant product after a single leucapheresis procedure and that the absence of concurrent lympholytic immunosuppression combined with a profoundly lymphopenic environment should allow for expansion and maintenance of the anti-CMV response in vivo.

This current study is a randomised prospective phase II study of pre-emptive adoptive cellular therapy for CMV following T cell depleted allogeneic HSCT from an unrelated donor. The study is based on earlier phase I-II studies of CMV-specific cellular therapy and our ongoing phase III study of CMV-specific adoptive cellular immunotherapy in immunocompromised recipients of allogeneic sibling donor HSCT based on selection of CMV-specific T cells by two different methodologies (CMV-IMPACT). The proof of safety in the sibling donor setting now strengthens the case for extending the therapy to the unrelated donor setting, where both potential risks and benefits are greater. The current study will investigate the use of CMV-specific T cells selected from mobilised blood collected at the time of stem cell apheresis by the multimer technology in the unrelated donor setting. The selection of CMV-specific T cells selected from a mobilised blood at the time of stem cell apheresis is in contrast to the methodology used in the CMV-IMPACT study where selection is performed on a non-mobilised blood product produced from a second study-dedicated apheresis. Two significant issues remain unresolved for the CMV-ACE/ASPECT study; are these infusions safe in the HLA-matched un-related donor setting and do CMV-reactive T cells derived from the transplant product have equivalent activity in vivo to cells derived from a second apheresis as used in the sibling donor study (CMV-IMPACT study). The study will test the hypothesis that ACT can augment the impaired CMV immune function post-transplant and reduce the requirement for CMV antiviral drug therapy without causing an increase in GVHD; and to determine the efficacy of pre-emptive CMV-specific adoptive cellular therapy following T cell depleted allogeneic HSCT with respect to reconstitution of CMV-reactive T cells. There are multiple methods for T cell depletion available, and differences between them will likely have an effect on immune reconstitution. The study will be restricted to patients receiving alemtuzumab-containing conditioning protocols, where the risk of CMV infection is greatest. ACT will be administered from day 21 post transplant for those receiving ex-vivo T-cell depleted grafts and day 28 for those receiving in vivo T cell depletion, as a single dose immediately upon a single CMV-DNA PCR+ result.

In summary the study is a multicentre, prospective, controlled, open label, randomised (2:1) study of pre-emptive infusion with CMV-specific T cells selected by the multimer selection technique plus standard CMV antiviral therapy versus standard CMV antiviral therapy alone.

The primary objective will be determine the efficacy of pre-emptive CMV-specific ACT following T cell depleted allogeneic HSCT with respect to reconstitution of CMV-reactive T cells and subsequent in vivo expansion of CMV-reactive T cells post infusion of ACT. In addition individual groups will be compared for duration of antiviral therapy and number of reactivation episodes, plus GVHD incidence.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16 years or older
2. cytomegalovirus seropositive allogeneic T cell depleted (alemtuzumab-containing conditioning regimen) hematopoietic stem cell transplant recipient with cytomegalovirus (CMV) seropositive unrelated donor
3. Patient Informed consent

   1. Prepared to undergo additional study procedures as per study schedule
   2. Patient has undergone counselling about risk
4. Donor engraftment (neutrophils > 0.5x109/l)(to be assessed prior to cytomegalovirus (CMV)-specific T cell infusion)
5. Single positive cytomegalovirus PCR result (And to be assessed prior to cytomegalovirus (CMV)-specific T cell infusion)
6. The donor will be selected from the Anthony Nolan Trust registry or other donor registries that have approved the protocol and consent procedure.
7. Donor must have met requirements of EU Tissue and Cells Directive(2004/23/EC) as amended and the UK statutory instruments pursuant therein.
8. Healthy, Cytomegalovirus (CMV)seropositive donor - having passed medical for stem cell donation
9. Subject and Donor must have negative serology for Human immunodeficiency virus (HIV), Hepatitis B and C, syphilis
10. human leukocyte antigen (HLA) type A*0101, A*0201, A*2402, B*0702 and B*0801
11. Donor informed consent for stem cell mobilisation leucapheresis and storage

Exclusion Criteria:

1. Pregnant or lactating women
2. Co-existing medical problems that would place the patient at significant risk of death due to Graft versus Host Disease (GVHD) or its sequelae
3. Human immunodeficiency virus infection
4. Active acute Graft versus Host Disease (GVHD) > Grade I (to be assessed prior to CMV-specific T cell infusion )
5. Concurrent use of systemic corticosteroids(to be assessed prior to cytomegalovirus (CMV)-specific T cell infusion )
6. Organ dysfunction (to be assessed prior to cytomegalovirus-specific T cell infusion ) as measured by:

   1. creatinine > 200 uM/l
   2. bilirubin > 50 uM/l
   3. alanine transferase > 3x upper limit of normal
7. Donor pregnant or lactating
8. Donor platelets < 50x109/l

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-10; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Cytomegalovirus (CMV) specific immune reconstitution | First two months
  Primary endpoint will be the peak number of circulating Cytomegalovirus (CMV)-reactive T cells within the first two months, after single positive cytomegalovirus PCR result (or post adoptive cell therapy infusion)

CONTACTS AND LOCATIONS:
Overall Officials: Karl S Peggs, Study Chair — University College London Hospital
Locations (9):
- United Kingdom (9):
  - QEH Birmingham Hospital, Birmingham
  - Bristol Royal Hospital, Bristol
  - University College London Hospital, London
  - Kings College Hospital, London
  - Royal Free Hospital, London
  - Manchester Royal Infirmary, Manchester
  - The Christie, Manchester
  - Nottingham University Hospital - City Campus, Nottingham
  - Churchill Hospital, Oxford